CLINICAL TRIAL: NCT02668367
Title: A Sequential-Cohort, Double-Blind, Placebo-Controlled, Multiple Ascending Oral Dose Study of the Safety and Pharmacokinetics of BTA-C585 in Healthy Volunteers
Brief Title: Safety and Pharmacokinetics Study of Multiple Ascending Doses of BTA-C585 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biota Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Vaxart (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTA585-002
Record Dates: First submitted 2016-01-27; First posted 2016-01-29 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Pharmacokinetics; Healthy Volunteers
Keywords: Viral Diseases; Antiviral; Paramyxoviridae Infections; RSV; Respiratory Syncytial Virus; Aviragen Therapeutics, Inc.; Aviragen Therapeutics; Aviragen
MeSH Terms: conditions — Virus Diseases; Paramyxoviridae Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BTA-C585 oral capsules (Active Comparator): 100 mg capsules; Multiple ascending doses (MAD) from 100 mg to 600 mg
  Interventions: Drug: BTA-C585 oral capsules
- BTA-C585 matching placebo (Placebo Comparator): BTA-C585 Matching placebo capsules; single doses
  Interventions: Drug: BTA-C585 matching placebo

INTERVENTIONS:
Drug: BTA-C585 oral capsules — BTA-C585; Multiple ascending doses from 100 mg to 600 mg
  Other Names: BTA585
  Arms: BTA-C585 oral capsules
Drug: BTA-C585 matching placebo — Multiple ascending doses to match 100 mg to 600 mg BTA-C585 capsules
  Other Names: BTA585
  Arms: BTA-C585 matching placebo

SUMMARY:
This is a single center, sequential-cohort, double-blind, placebo-controlled, multiple ascending dose (MAD), 7-day treatment period study in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women;
2. Age 18 to 60 years, inclusive;
3. Weight ≥ 50 kg and Body Mass Index (BMI) of 19 to 32, inclusive;
4. Female subjects must be of non-childbearing potential;
5. Male subjects must agree to use a double barrier method of birth control;
6. Signed informed consent form (ICF) prior to study procedures.

Exclusion Criteria:

1. Current or recent (within 14 days of Day 0) bacterial or viral infection;
2. Positive results at screening for hepatitis B surface antigen, hepatitis C antibody, or HIV antibody;
3. Clinically significant abnormalities noted on ECG;
4. Safety laboratory abnormalities;
5. Regular use of medications, prescription or non-prescription;
6. Poor vein access or fear of venipuncture or sight of blood;
7. Major surgery, significant recent injury or trauma within 30 days;
8. Received an investigational drug or vaccine within 30 days.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) from time 0 to 24 hours | 0-24 hours
Number of adverse events | Day -1 to Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Anna Novotney-Barry, Study Director — Biota Pharmaceuticals, Inc.
Locations (1):
- Biota Investigational Site, San Antonio, Texas, United States